CLINICAL TRIAL: NCT02622399
Title: Mobilizing Community Networks to Optimize Child Well-being
Acronym: NOW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Principal Investigator, Renee Boynton-Jarrett, BMC Attending Physician, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: H-33938
Record Dates: First submitted 2015-11-16; First posted 2015-12-04 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Social Isolation
MeSH Terms: conditions — Social Isolation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Project NOW (Experimental): Participants in the intervention arm receive access to free mobile communications and a web-based informational platform supported by txtwire.
  Interventions: Behavioral: Project NOW
- Control (No Intervention): Participants in the control arm do not receive access to the txtwire platform.

INTERVENTIONS:
Behavioral: Project NOW — This intervention aims to reduce social isolation and promote engagement in health promoting enrichment and activities, by embedding a community health worker-assisted forum in a community-driven mobile communications through a private, secure, and confidential platform supported by txtwire. The principal innovation is harnessing both the behavioral change utility of a mobile health application and the social support potential of an online social network the investigators can deliver more timely and dynamic reinforcement to caregivers and social support more in rhythm with the pace of community events and stressors.
  Arms: Project NOW

SUMMARY:
Caregiver social isolation adversely impacts child health and developmental outcomes; it also contributes to suboptimal engagement in health care services and enrichment resources, which also elevate risk for poor outcomes in childhood. The proposed pilot intervention aims to reduce social isolation and promote engagement in health promoting enrichment and activities, by embedding a community health worker assisted forum in a community-driven mobile communications (using a platform supported by the company txtwire).

The investigators propose a two-arm, pilot study enrolling 100 parents of children age 0-5 years old who reside in the Roxbury, Dorchester, and Mattapan neighborhoods of Boston. Participants will be recruited from Boston Medical Center and community sites in Roxbury, Dorchester, and Mattapan. The investigators will use quality improvement methods to improve the utilization of the mobile communications shared through txtwire to build collective efficacy for children and social support and engagement that will optimize family resiliency and thereby promote child well-being, as well as, assess the acceptability of the intervention, and logistics of the field implementation to ultimately inform an appropriately powered RCT. Participants will receive compensation for participation at baseline and follow-up interviews.

The intent of this study is to support developement of mobile social communications to reduce social isolation.

DETAILED DESCRIPTION:
The investigators propose a two-arm, pilot study enrolling 100 parents of children age 0-5 years old who reside in the Dudley Square neighborhood of Boston. Participants will be recruited from Boston Medical Center and community sites in Dudley Square. After completing the baseline survey, 50% of participants will be randomized to receive access to a free mobile communications and a web-based informational platform supported by txtwire. A simple randomization technique will be used.

The investigators will engage a group of community residents (who are not study participants) in the process of designing the social network content for the txtwire site and features.

The investigators will use quality improvement methods to improve the utilization of the txtwire mobile communications to improve social support and engagement that will optimize family resiliency and thereby promote child well-being, as well as, assess the acceptability of the intervention, and logistics of the field implementation to ultimately inform an appropriately powered RCT.

Recruitment will take place at Boston Medical Center in the outpatient pediatric primary care clinic and at public, community sites in Dorchester, Roxbury and Mattapan. The investigators will have a trained research assistant approach and recruit parents who are presenting for well-child care visits. The locations will be selected to maximize convenience for the families. A trained research assistant, following this standard procedure will screen parents presenting with a child between the ages of 0 and 5 years old for a routine health care maintenance visit from the clinical waiting areas at BMC and from public community sites.

Participants will be approached by a trained research assistant who will share a 1-page flyer about the study (see attached) and ask if they would like to proceed with the eligibility screening. For patients who meet inclusion/exclusion criteria, formal consent and contact information will be obtained. In order to proceed with the interview parents must agree to a follow-up interview in 6-months via phone or in-person.

Participants will be approached in the clinic waiting area at Boston Medical Center and in open community sites in the Dorchester, Roxbury, and Mattapan neighborhoods.

1. First, the investigators will conduct a preliminary eligibility screen to determine participant eligibility using the criteria described below.
2. Next, each participant will complete a contact information form that includes name, cell phone number, home address, and email address.
3. Next, Each participant will complete a baseline survey.

After completing the baseline survey, the investigators will randomize 50% of participants to the intervention arm: the free txtwire social mobile communications. The investigators will randomize 100 caregivers with a child between the ages of 0-5 years old and have a primary residence in the Dorchester, Roxbury, or Mattapan neighborhoods of Boston. 50% of participants will be randomized to the free txtwire mobile communications. With the exception of cellphone number there will be no identifying data recorded by txtwire.

Subjects will be randomly allocated to study arms to eliminate unmeasured confounding. For those who consent, the investigators will randomize 1:1, according to a pre-made, concealed schedule. Subjects will be randomized to txtwire mobile communications or no intervention. Fifty caregivers in the intervention arm will receive a brief, in-person, training on how to use the txtwire mobile communications and assistance with setting it up on their mobile devices. Fifty caregivers will be randomized to the control arm. Members of the control arm will not receive any additional training or app. For both arms, the investigators will track engagement with community resources and services for child health and enrichment, social support and networks, and child and family well-being over a 6 month period using brief monthly electronic surveys completed on the mobile phone. These surveys will be administered using Mobile Commons. At the end of the 6 month period all subjects will complete a follow-up survey. They will receive compensation for completion. If an in-person interview is not possible, the investigators will conduct a phone interview.

The investigators will meet with community members who are not study participants to receive feedback on the content, layout, txtwire platform.

The investigators will meet biweekly as a team with the Community Health Worker, Research Assistant, Dr. Boynton-Jarrett and data manager. Using the Institute for Healthcare Improvement's Model for Improvement Plan-Do-Study-Act (PDSA) methodology, the investigators will review the use of the txtwire mobile communications and attempt to improve functioning of the community health worker mediated forum in an iterative fashion. Intervention study participants will be able to provide feedback on the utility of information provided through the txtwire mobile communications using the online platform. The investigators will plan for a change in one facet of the intervention, implement that change (do), study whether the desired effect was achieved, and act to determine if further optimization is needed. The investigators hope to engage in two or three PDSA cycles during the intervention period.

The investigators will conduct a semi-structured qualitative interviews with our intervention subjects to better understand engagement with the txtwire mobile communications at the time of the follow-up survey. The investigators intend to use the qualitative interview techniques to understand attitudes, behaviors, and motivations for interacting with the system.

ELIGIBILITY:
Inclusion Criteria:

* Must be a parent or primary caregiver for child five years or younger
* Participant has a smart phone that is text message and web enabled
* Participant resides in the Dorchester, Mattapan, or Roxbury neighborhoods of Boston, within the 02119, 02121, 02122, 02124, 02125, 02126 zip codes
* Fluent in English language
* Able to participate in English.

Exclusion Criteria:

* Does not have a smart phone or the ability to navigate a mobile application
* Participant does not reside Dorchester, Mattapan, or Roxbury neighborhoods of Boston, within the 02119, 02121, 02122, 02124, 02125, 02126 zip codes
* Not identified as a parent or caregiver of a child age five years old or younger
* Not identified as a parent or caregiver of a child age five years old or younger

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 98 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Reduction in social isolation | 6 months
  This will be measured by change in baseline to follow-up survey on measures of social isolation.

SECONDARY OUTCOMES:
Decrease in parental stress | 6 months
  These will be obtained via self-report and assessment of change between the baseline and follow-up survey.
Increase in parental social support | 6 months
  These will be obtained via self-report and assessment of change between the baseline and follow-up survey.
increase in parental knowledge of and use of community resources for child enrichment and well-being | 6 months
  These will be obtained via self-report and assessment of change between the baseline and follow-up survey.

CONTACTS AND LOCATIONS:
Overall Officials: Renee Boynton-Jarrett, MD, ScD, Principal Investigator — Associate Professor
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No